CLINICAL TRIAL: NCT02749643
Title: The Effects of Adding Vibrotactile Feedback to Prostheses on Functional Outcome Measures of Transradial Amputation Prosthetic Users
Brief Title: Functional Outcome Measures With Vibrotactile Feedback to Prostheses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Isabella Shvartz, Director, clinical research, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VTF- HMO-CTIL
Record Dates: First submitted 2016-04-13; First posted 2016-04-25 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Unilateral Transradial Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vibrotactile feedback (Experimental): Vibrotactile system - comprises of force sensors, attached to the fingertips of the prosthetic hand, and a set of 8 vibration actuators attached to a fabric arm cuff. When the subject applies force on the sensors with his prosthetic hand, he receives a vibration on the skin of his arm. The sensors and actuators are connected to an electronic control board, which transforms the resistance from the sensors to an electric signal that activates the vibration actuators.
  Interventions: Device: Vibrotactile feedback system

INTERVENTIONS:
Device: Vibrotactile feedback system

SUMMARY:
Investigators wish to evaluate the effects of adding VTF to upper limb prostheses on functional outcome measures of upper limb prosthetic users.

DETAILED DESCRIPTION:
Investigators will perform three experiments:

1. Investigators will add vibrotactile feedback to prosthetic users during the execution of a standardized functional test and performance of simple grasping tasks, with a disruption to the normal visual feedback, and examine whether their performance and arm kinematics are improved with tactile feedback;
2. Investigators will examine the effects of adding the feedback to a prosthesis on the performance and visual attention during a dual task assignment in prosthetic users, and
3. Investigators will provide prosthetic users with the feedback, to use it at their natural surroundings for a week, and study the reported activity and satisfaction levels.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transradial amputee
* Using a transradial myoelectric prosthesis
* Ability to follow simple instructions, understand and sign an informed consent form
* Normal or corrected eyesight

Exclusion Criteria:

* Elbow or wrist disarticulation or partial hand amputations
* Neuropathy or skin ulcers on the amputated limb

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Orthotics and Prosthetics User Survey-Upper Extremity Functional Status | 2 weeks
  A subjective questionnaire concerning the ability to perform daily tasks. The score ranges from 23 to 115.

SECONDARY OUTCOMES:
Modified Box & Blocks test | 2 weeks
  This test is aimed to assess unilateral gross manual dexterity. The test comprises of a two-compartment box and 16 cube blocks.The subject is instructed to transport the blocks as possible over the partition into the opposite compartment. The time in seconds is measured.
Time to complete dual tasking test | 2 weeks
  The time needed to complete grasping tasks while playing a simple computer game with the other hand is measured in seconds.
Activity | 2 weeks
  In order to record the actual use of the prosthesis in the natural environment of the subject, a wireless activity monitor that can be easily attached to the prosthesis will be used. The output measure of the activity monitor are "activity counts".

CONTACTS AND LOCATIONS:
Overall Officials: Sigal Portnoy, PhD, Study Director — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Clemente F, D'Alonzo M, Controzzi M, Edin BB, Cipriani C. Non-Invasive, Temporally Discrete Feedback of Object Contact and Release Improves Grasp Control of Closed-Loop Myoelectric Transradial Prostheses. IEEE Trans Neural Syst Rehabil Eng. 2016 Dec;24(12):1314-1322. doi: 10.1109/TNSRE.2015.2500586. Epub 2015 Nov 13. PMID 26584497
- [Derived] Raveh E, Portnoy S, Friedman J. Myoelectric Prosthesis Users Improve Performance Time and Accuracy Using Vibrotactile Feedback When Visual Feedback Is Disturbed. Arch Phys Med Rehabil. 2018 Nov;99(11):2263-2270. doi: 10.1016/j.apmr.2018.05.019. Epub 2018 Jun 20. PMID 29935153